CLINICAL TRIAL: NCT04000061
Title: Heart Failure-USB: Prediction and Progression
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-00956; me19Mueller
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Acute Heart Failure; Acute Coronary Syndrome; Heart Failure
MeSH Terms: conditions — Acute Coronary Syndrome; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- acute coronary syndrome (ACS): Outcome information (all-cause death, heart failure (HF) hospitalizations) of patients hospitalized with a primary diagnosis of ACS is analyzed.
  Interventions: Other: medical chart review; Other: data generated by direct IT export
- acute heart failure (AHF): Outcome information (all-cause death, heart failure (HF) hospitalizations) of patients hospitalized with a primary or secondary diagnosis of AHF is analyzed.
  Interventions: Other: medical chart review; Other: data generated by direct IT export

INTERVENTIONS:
Other: medical chart review — data generated by medical review include Medical history, Medications at presentation, during hospitalization and at discharge, New York Heart Association (NYHA) class, Killip class, Electrocardiographic (ECG) data, echocardiographic data, Interventions (Percutaneous Coronary Intervention (PCI), Coronary Artery Bypass Graft (CABG), Implantable Cardioverter Defibrillator (ICD) implantation, Cardiac Resynchronization Therapy (CRT) Implantation), Outcome Information: all-cause death, HF hospitalizations
Other: data generated by direct IT export — data generated by direct IT export include Anthropometric data (age, sex, height, weight), Vital signs, Laboratory data

SUMMARY:
This retrospective cohort study is to identify triggers of heart failure (HF) development and drivers of HF progression as well as the underlying cardiac disease (phenotype) to identify patients at risk and predict the clinical course of the disease. Data of patients who were hospitalized during the years 2010-2023 with acute coronary syndrome (ACS) and/ or with acute heart failure (AHF) will be collected and analyzed. In a subgroup cohort efficacy and safety of digoxin in patients with acute heart failure triggered by tachyarrhythmia will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized with a primary diagnosis of ACS
* Patients hospitalized with a primary or secondary diagnosis of AHF

Exclusion Criteria:

* Existence of a documented statement of the patient against the scientific use of clinical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that were hospitalized at the Universitätsspital Basel/ Switzerland with the diagnosis of ACS or AHF during the years 2010 - 2023
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2019-06-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
number of all-cause death | 1 to 8 years after hospitalization
  number of all-cause death in patients hospitalized with ACS and AHF during the years 2010-2023.
number of HF hospitalizations | 1 to 8 years after hospitalization
  number of new HF hospitalizations in patients hospitalized with ACS and AHF during the years 2010-2023
number of cardiovascular death | 1 to 8 years after hospitalization
  number of cardiovascular death in patients hospitalized with ACS and AHF
number of cardiovascular hospitalizations | 1 to 8 years after hospitalization
  number of cardiovascular hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Christian Müller, Prof. Dr., Principal Investigator — Cardiology University Hospital Basel
Locations (1):
- Cardiology, University Hospital Basel, Basel, Switzerland